CLINICAL TRIAL: NCT07163936
Title: Analysis of the Influence of Dialysis Fluid Composition on Vascular Calcification in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Acronym: CalCio-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2024/0318
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Vascular Calcification; Hemodialysis; Cardiovascular Disease (CKD)
Keywords: hemodialysis; dialysate; citrate dialysate; acetate dialysate; magnesium supplementation; calcification propensity; vascular calcification; dialysate composition
MeSH Terms: conditions — Vascular Calcification; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label, single-center clinical trial with 12 months of follow-up. Participants will be randomly assigned in a 1:1 ratio to one of two study arms:
  Control group: Hemodialysis with acetate-based dialysate (Fresenius SmartBag 211.5)
  Intervention group: Hemodialysis with citrate-based dialysate containing magnesium supplementation (Fresenius SmartBag CA 211.5-0.75)
  Both dialysates are routinely used in clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetate dialysate (Active Comparator): Fresenius SmartBag 211.5
  Interventions: Device: Acetate dialysate
- Citrate dialysate (Experimental): Fresenius SmartBag CA 211.5-0.75
  Interventions: Device: Citrate dialysate with magensium supplementation

INTERVENTIONS:
Device: Citrate dialysate with magensium supplementation — Citrate-based bicarbonate dialysate containing: sodium 138 mmol/L, chloride 110 mmol/L, potassium 2 mmol/L, calcium 1.5 mmol/L, magnesium 0.75 mmol/L, citrate 1 mmol/L, glucose 1 g/L, bicarbonate 32 mmol/L.
  Arms: Citrate dialysate
Device: Acetate dialysate — Acetate-based bicarbonate dialysate containing: sodium 138 mmol/L, chloride 109 mmol/L, potassium 2 mmol/L, calcium 1.5 mmol/L, magnesium 0.5 mmol/L, acetate 3 mmol/L, glucose 1 g/L, bicarbonate 32 mmol/L.
  Arms: Acetate dialysate

SUMMARY:
The goal of this clinical trial is to find out if using a citrate-based dialysate with added magnesium during hemodialysis can help slow down or prevent the hardening of blood vessels (vascular calcification) in adults on long-term dialysis.

The main questions the study will try to answer are:

Does citrate-based dialysate with magnesium improve the blood's ability to prevent calcium buildup (measured by a test called T50) compared to acetate-based dialysate?

Does it modify magnesium, calcium and parathyroid hormone (PTH) levels in the blood?

Does it lower the chances of heart problems or death?

Researchers will compare two groups: one will receive acetate-based dialysate, and the other will receive citrate-based dialysate with magnesium.

Participants will:

Receive one of the two types of dialysate during their regular hemodialysis sessions for 12 months

Have regular blood tests

Be monitored for any heart problems and for overall health during the study

DETAILED DESCRIPTION:
Vascular calcification is a common and serious complication in patients receiving long-term hemodialysis. Dialysate composition may influence its progression. Acetate, a weak acid, has traditionally been added to dialysate to maintain chemical stability and prevent precipitation of calcium or magnesium bicarbonate salts. However, long-term acetate exposure has been associated with adverse effects, prompting the search for safer alternatives.

Citrate is a promising substitute that may help reduce vascular calcification by maintaining a neutral calcium balance. Nevertheless, it can lower magnesium levels in the blood (hypomagnesemia), which might counteract its benefits. This supports the idea of adding magnesium to citrate-based dialysate.

This is a prospective, randomized, open-label clinical trial designed to compare the effects of acetate-based dialysate versus citrate-based dialysate with magnesium supplementation in adult hemodialysis patients. Participants will be enrolled and followed for 12 months.

The primary outcome will be changes in calcification propensity (T50). Secondary outcomes include changes in serum magnesium, calcium, and PTH levels, as well as the incidence of cardiovascular events and all-cause mortality.

The findings may help identify a safer and more effective dialysate composition to improve cardiovascular outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) on maintenance hemodialysis for more than 3 months
* Clinically stable patients with a well-functioning vascular access
* Residual urine output ≤ 250 mL/day
* Able and willing to provide written informed consent

Exclusion Criteria:

* Known allergy or intolerance to any component of the dialysates
* Active malignancy or infectious/inflammatory disease
* Planned living donor kidney transplant before study completion
* Current treatment with vitamin K antagonists (coumarins)
* Severe hypocalcemia or poorly controlled secondary hyperparathyroidism
* Any condition that, in the investigator's judgment, contraindicates participation or affects study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2026-09-06 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
Calcification propensity (T50 test) | Baseline and at 3, 6, 9, and 12 months
  T50 is a laboratory test that measures the serum's intrinsic capacity to inhibit calcium-phosphate precipitation, reflecting the overall propensity for vascular and soft tissue calcification. Higher T50 values indicate greater calcification resistance.

SECONDARY OUTCOMES:
Serum magnesium levels | Baseline and at 3, 6, 9, and 12 months
  Measurement of total serum magnesium to assess electrolyte balance and detect hypomagnesemia or hypermagnesemia during the intervention.
Total serum calcium levels | Baseline and at 3, 6, 9, and 12 months
  Measurement of total calcium to monitor mineral metabolism and calcium homeostasis.
Parathyroid hormone (PTH) levels | Baseline and at 3, 6, 9, and 12 months
  Measurement of intact parathyroid hormone to assess bone-mineral metabolism and response to dialysate composition.
Serum vitamin D levels | Baseline and at 3, 6, 9, and 12 months
  Measurement of serum 25-hydroxyvitamin D to evaluate vitamin D status and its potential influence on mineral metabolism.

OTHER OUTCOMES:
Cardiovascular events and all-cause mortality | During the 12-month follow-up period
  Number and type of cardiovascular events, including myocardial infarction, stroke, heart failure, and hospitalization due to cardiovascular causes, as well as number of deaths from any cause during the study period.

IPD SHARING:
Plan to Share IPD: Yes
IPD including de-identified laboratory results, demographic and clinical variables, and primary and secondary outcome data will be shared. Data will be anonymized to protect patient confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting from the date of study results publication and will remain accessible indefinitely.
Access Criteria: De-identified individual participant data and supporting documents will be made publicly available on a GitHub repository. Researchers and the public can access and download the data freely without restriction. Data will be anonymized to protect participant confidentiality. Users will be encouraged to cite the original study when using the data.